CLINICAL TRIAL: NCT02933125
Title: Effectiveness of Family-based Group Psychotherapy for Adolescents With Illicit Drug Use
Brief Title: Group Psychotherapy for Adolescents With Substance Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104-1729C
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2013-06

CONDITIONS: Substance Abuse
Keywords: substance abuse; group psychotherapy; family therapy; longitudinal study; child and adolescent
MeSH Terms: conditions — Substance-Related Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The youths in the intervention group will participate in a weekly 10-session out-patient motivational enhancement psychotherapy (MEP) program. In addition to this, these youths' caregivers will be referred to simultaneously take part in a weekly 10-session out-patient parenting skill training (PST) program at Kaohsiung Chang Gung Memorial Hospital.
  Interventions: Behavioral: Group psychotherapy
- Comparison group (Active Comparator): The comparison group consists of substance-using adolescents that receive only standard supervision by the protection officers in Taiwan's Kaohsiung Juvenile and Family Court. The protection officers provide the adolescents with moral education, as well as counseling in their work or studies.
  Interventions: Behavioral: Standard supervision

INTERVENTIONS:
Behavioral: Group psychotherapy — Motivational enhancement psychotherapy (MEP) for Youths:
  The participating youths have to attend one session a week for 10 weeks of a group program for relapse prevention based on motivational enhancement ideas and led by two experienced psychologists from the hospital.
  Parenting skill training (PST) for Caregivers:
  The PST program for the youths' caregivers also consist of 10 weekly, 120-minute sessions that were led by a senior consulting psychologist.
  Arms: Intervention group
Behavioral: Standard supervision — The standard supervision by the protection officers in Taiwan's Kaohsiung Juvenile and Family Court provide the adolescents with moral education, as well as counseling in their work or studies.
  Arms: Comparison group

SUMMARY:
Background: Substance abuse among children and adolescents is an important public health issue in Taiwan. Kaoshiung Chang Gung Memorial Hospital and Taiwan Kaoshiung Juvenile and Family Court will cooperate in a counseling program for adolescents with illicit drug abusers in 2013, to perform a mandatory 10-week family-based group psychotherapy.

Aims: This study aims (1) to investigate the effectiveness of the family-based group psychotherapy for adolescents with illicit drug abusers and their parents; (2) to identify whether the counseling program is effective for preventing the adolescents from relapse of substance abuse.

Expected Results: The investigators expect that (1) group psychotherapy may involve comprehensive benefits for adolescents with illicit drug abusers, by improving the changes in adolescents' substance-craving symptoms and behavioral problems, and reducing stress of their parents; (2) this counseling program is effective for preventing the adolescents from relapse of substance abuse; (3) the findings in this study will not only demonstrate empirical evidence of treatment effectiveness for adolescents with illicit drug abuse, but will also provide useful clues for future implementation of policy making.

DETAILED DESCRIPTION:
1. The investigators plan to recruit 200 adolescents (=< 20 years) with illicit drug abusers and their parents (100 of intervention group and 100 of comparison group).
2. The intervention group consists of youths that participate in a program that combines a weekly 10-session out-patient motivational enhancement psychotherapy (MEP) program for youths with an additional weekly 10-session parenting skill training (PST) program for their guardians.
3. The comparison group consists of youths that receive standard supervision by the court. All participants were followed up for a maximum of three years.
4. The assessments for adolescents and their parents will be taken at pre- and post-treatment, using the Adolescents' Behavior-problem Scale, the Craving Beliefs Questionnaire, the Family APGAR, the Parenting Stress Index-Short From (PSI/SF) and the Chinese Health Questionnaire (CHQ).
5. The information of adolescents' relapse of substance abuse will be collected by Kaoshiung Juvenile and Family Court.

ELIGIBILITY:
Inclusion Criteria:

* The adolescents with illicit drug age between 12 to 20.
* One of their parents can attend the counseling program.

Exclusion Criteria:

* The adolescents or their parents can't attend the program.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Substance-use relapse | Longitudinal follow-up for 3 years
  Relapse is defined as positive urine test for any substance within the follow-up period.
Academic or social status | Longitudinal follow-up for 3 years
  The academic or social outcome is categorized into as attending school, being employed, or being a dropout/unemployed.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, MD, MPH, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No